CLINICAL TRIAL: NCT04564859
Title: The Efficiency of Heated Humidifier High-Flow Nasal Cannula Between Unheated Oxygen Therapy in Difficult Weaning Patients After Extubation in Respiratory Care Center
Brief Title: The Efficiency of HHHFNC Between Unheated Oxygen Therapy in Difficult Weaning Patients After Extubation in RCC
Acronym: HHHFNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Collaborators: Fu Jen Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SKH-8302-106-NDR-05
Record Dates: First submitted 2020-09-13; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Critically Illness
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noninvasive Ventilation group (Experimental): Noninvasive Ventilation group initial setting： Insp. Pressure：12 ~ 16 centimeter of water Exp. Pressure ： 4 ~ 6 centimeter of water FiO2：Keep oxygen saturation measured by pulse oximeter：> 92% By condition, gradually tap 2~3 centimeter of water inspiratory positive airway pressure Keep Tidal volume：6~10 ml/kg
  Interventions: Device: Heated Humidified High-Flow Nasal Cannula
- Heated Humidified High-Flow Nasal Cannula group (Active Comparator): Heated Humidified High-Flow Nasal Cannula group initial setting： Flow setting: 50 L/m FiO2：Keep oxygen saturation measured by pulse oximeter > 92% temperature:37 ℃ By condition, gradually tap Flow 5 L/m
  Interventions: Device: Heated Humidified High-Flow Nasal Cannula

INTERVENTIONS:
Device: Heated Humidified High-Flow Nasal Cannula — Participants using of invasive ventilator more than 14 days, maybe considered transferred to the Respiratory Care Center(RCC), participants enrolled to this study and also written informed consent from participants or their family; After extubation, the difficult weaning patients were allocated to two treatment groups, and randomly assigned to Heated Humidified High-Flow Nasal Cannula or Noninvasive Ventilation devices.
  Other Names: Noninvasive Ventilation

SUMMARY:
The purpose of this study is to assess the efficacy of Heated Humidified High-Flow Nasal Cannula compared with noninvasive positive-pressure ventilation in the prevention of extubation failure in patients with prolonged mechanical ventilation.

DETAILED DESCRIPTION:
There have been many clinical trials comparing the role of Heated Humidified High-Flow Nasal Cannula or Noninvasive positive pressure ventilation in the prevention of extubation failure.

These review all have similar results summarized here:

Compared with Noninvasive positive pressure ventilation, Heated Humidified High-Flow Nasal Cannula provides better patient comfort, fewer oxygen desaturation episodes, lower likelihood of interface displacement, and, lower reintubation rate than Noninvasive positive pressure ventilation.

However, most of these clinical trials focused on participants experiencing acute respiratory failure.

Investigators of this study want to find something difference between oh these two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: Over 20 years of age
* the requirement of at least six hours of mechanical ventilation per day for at least 14 consecutive days

Exclusion Criteria:

* Pregnancy
* Status post tracheostomy
* Neuromuscular diseases
* Signed "do not resuscitate" order
* Unplanned extubation

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Re-intubation rate | within 72 hours of extubation
  Any placement of an endotracheal tube for any indication within 72 hours of extubation, censored at the first of hospital discharge or 72 hours after extubation.

SECONDARY OUTCOMES:
Mortality rate | up to 3 months
  Mortality rate, or death rate is a measure of the number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Chun Lin, MD, Study Chair — Shin Kong Wu Ho-Su Memorial Hospital

REFERENCES:
- [Derived] Tseng CW, Chao KY, Wu HL, Lin CC, Hsu HS. Effectiveness of high-flow nasal cannulae compared with noninvasive positive-pressure ventilation in preventing reintubation in patients receiving prolonged mechanical ventilation. Sci Rep. 2023 Mar 22;13(1):4689. doi: 10.1038/s41598-023-31444-8. PMID 36949116